CLINICAL TRIAL: NCT07130487
Title: Project CARE: CAncer Risk Evaluation (CARE)
Brief Title: Project CARE: CAncer Risk Evaluation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anita Y. Kinney, PhD, RN (Other)
Responsible Party: Sponsor-Investigator, Anita Y. Kinney, PhD, RN, Director at Rutgers Cancer Institute, Rutgers, The State University of New Jersey
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: Pro2024002233
Record Dates: First submitted 2025-07-31; First posted 2025-08-19 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Primary Care
Keywords: Genetic Counseling; Genetic Testing; Primary Care Provider; High-risk patients in primary care settings; Genetic Education; Relational Agent; Chatbot
MeSH Terms: interventions — Darbepoetin alfa

STUDY DESIGN:
Intervention Model Description: This single-arm study intervention is Alex , a proactive digital relational agent developed through community participatory research and user-centered design. It provides interactive, literacy-conscious content that simulates traditional hereditary cancer risk assessment. High-risk patients, once identified, receive genetic education and counseling (GC), enabling direct access to genetic testing (GT) after engaging with the platform. Alex is HIPAA-compliant and aligned with NCCN guidelines. The chatbot evaluates patient-reported personal and family history to determine hereditary cancer GT eligibility. Its clinical content was designed by ABGC-certified genetic counselors (with expertise in hereditary cancer syndromes), behavioral scientists, and an epidemiologist.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Feasibility and Acceptability of Relational Agent Chatbot (Experimental)
  Interventions: Behavioral: Relational Agent ( RA) Alex

INTERVENTIONS:
Behavioral: Relational Agent ( RA) Alex — The intervention is an RA (chatbot) integrated into a genetic care delivery portal for primary care patients. The RA provides hereditary cancer education and risk evaluation through an interactive interface. Primary care patients will use the RA to complete questionnaires about their hereditary cancer risk, track their progress through the education component and assessment process, and obtain downloadable summaries of their cancer risk and family tree. Additionally, the chat feature stores past conversations, and a menu guides participants through key steps.

SUMMARY:
The purpose of Project CARE (cancer risk assessment and evaluation) research study is to explore the acceptance and feasibility of a study-initiated proactive outreach and digital care delivery model for conducting hereditary cancer risk assessment in primary care settings and facilitating genetic risk evaluation for patients flagged as high risk. Potential participants will be recruited from Rutgers Health primary care sites (family practice and general internal medicine). EPIC will be used to identify all potential participants and they will be invited to participate in the study. Consented participants will be provided a link via email, and or text message to engage with a Relational Agent (RA, chatbot), through the patient portal for cancer risk assessment and genetic education. Those identified as high risk will be offered genetic counseling and testing.

The research questions the study aims to answer are:

1. What percent of patients who completed the RA are identified as high risk?
2. What percent of patients who engaged with the risk assessment were identified as high risk?
3. What percent of high-risk patients had genetic counseling or genetic testing within 4 months of completing the risk assessment?

ELIGIBILITY:
Inclusion Criteria

1. Age 18 to 70 years
2. Able to read and speak English
3. Have an email address or mobile phone number in EPIC and/or are enrolled in MyChart
4. Receiving health care in Family Medicine or General Internal Medicine at Rutgers Health within the past 2 years
5. Have not opted out of receiving research-related communications
6. Have internet access (via smartphone, tablet, or computer)

Exclusion Criteria

1. Dementia (e.g., Alzheimer's disease) as indicated in EPIC
2. Unable to access the Internet (via smartphone, tablet, or computer)
3. Previous germline genetic testing for hereditary cancer risk
4. Opted out of research participation in EPIC
5. Have a personal history of cancer

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2025-11-19 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Proportion of Patients Completing the Hereditary Cancer Risk Assessment | Up to 3 months from enrollment
  The proportion of patients who successfully complete the hereditary cancer risk assessment within the genetic care delivery portal. Completion is defined as receiving a final result statement, regardless of whether all assessment questions in the risk assessment module were answered.
Proportion of Patients Identified as High Risk | Through study completion, an average of 12 months.
  The percent of patients who completed the RA and are identified as high risk.

SECONDARY OUTCOMES:
RA Engagement Rate | Up to 3 months from enrollment
  The number of patients invited to participate in the study who engaged with the RA link by clicking on the introductory response, divided by the total number of patients invited to the study, multiplied by 100.
Retention Rate of High-risk Participants at 1-Month | 1-month post high-risk identification
  The number of high-risk participants who complete the 1-month follow-up survey divided by the number of high-risk participants, multiplied by 100.
Satisfaction with the Risk Assessment Feature of the Relational Agent | Through study completion, an average of 12 months.
  Participant satisfaction will be assessed using a two-item questionnaire (Relational Agent Satisfaction Scale, adapted), with each item rated on a 1-5 scale (1 = very dissatisfied; 5 = very satisfied). Higher scores indicate greater satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Anita Y Kinney, PhD, RN, Principal Investigator — Rutgers, The State University of New Jersey
Locations (1):
- Rutgers, The State University of New Jersey, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will not be shared due to privacy concerns and to protect participants' confidentiality.